CLINICAL TRIAL: NCT00014898
Title: Attention Deficit Disorder and Exposure to Lead
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 5015-CP-001
Record Dates: First submitted 2001-04-12; First posted 2001-04-13 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Attention Deficit Disorder
Keywords: Lead exposure; Bone lead; Attention deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
We are examining the past exposure to lead in 250 well characterized children with ADHD, and a suitable group of controls. Our measure of past exposure is bone lead levels obtained by XRay fluorescence spectroscopy, a relatively new way of estimating bone lead concentrations, and by inference, body lead burdens. By comparing the lead concentrations in these two groups, controlling for other factors which could confound, we will estimate odds ratios for ADHD given elevated bone lead, and estimate the contribution of lead to this disease of childhood.

ELIGIBILITY:
Case subjects are drawn from adolescents aged 10 to 18 previously seen at Western Psychiatric Institute and Clinic for evaluation, and meet the DSM-IIIR criteria for diagnosis of ADHD based on a structured parent interview and standardized parent and teacher rating scales. Cases were also systematically observed and evaluated in the summer treatment program between 1987 and 1996 at WPIC. Controls are demographically matched non-ADHD adolescents, recruited from surrounding communities and pediatric practices.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500
Dates: Start 1999-06; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States